CLINICAL TRIAL: NCT02563990
Title: The Impact of Injection Pressure During Adductor Canal Nerve Block
Brief Title: Injection Pressure & Adductor Canal Block
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit additional patients due to transfer of surgical service (ortho sports medicine) and recruitable cases to another institution.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Andres Missair, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20150583
Record Dates: First submitted 2015-09-25; First posted 2015-09-30 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Orthopedic Disorders; Injury of Anterior Cruciate Ligament
MeSH Terms: conditions — Musculoskeletal Diseases; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Pressure (Experimental): High pressure injection of Ropivacaine local anesthetic at greater than 20 psi
  Interventions: Procedure: High Pressure Injection
- Low Pressure (Active Comparator): Low pressure injection of Ropivacaine local anesthetic at less than 15 psi
  Interventions: Procedure: Low Pressure Injection

INTERVENTIONS:
Procedure: High Pressure Injection — Adductor canal block performed at greater than 20 psi injection pressure
  Arms: High Pressure
Procedure: Low Pressure Injection — Adductor canal block performed at less than 15 psi injection pressure
  Arms: Low Pressure

SUMMARY:
This is a prospective, randomized, single-blinded human clinical trial that will examine how injection pressure influences the spread of a given volume of injectate in the adductor canal, during adductor canal nerve block.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blinded human clinical trial that will examine how injection pressure influences the spread of a given volume of injectate in the adductor canal, during adductor canal nerve block. The study population will be patients undergoing elective anterior cruciate ligament repair in the distal lower extremity and receiving preoperative adductor canal nerve blocks for postoperative analgesia. They will be randomized into two groups of 25 patients each. The investigators speculate that high injection pressures (>20 psi) will lead to greater spread of local anesthetic than low injection pressures (<15 psi) during mid-thigh adductor canal nerve blocks. The primary endpoint is the spread of injectate, defined as the distance between the uppermost and lowermost limits of spread of local anesthetic as assessed by ultrasound. The secondary endpoints are the incidence of femoral and sciatic nerve blocks 30 minutes after block placement, amount of IV opioid administered intraoperatively and postoperatively, preoperative and postoperative pain (Numeric Rating Scale, 0-10), and postoperative physical therapy milestone achievement.

ELIGIBILITY:
Inclusion criteria:

1. Planned general anesthetic.
2. American Society of Anesthesia classes I, II, or III.
3. Patients aged 18-65.
4. English-speaking patients.

Exclusion criteria:

1. ASA classes IV and V.
2. Patients younger than 18 or older than 65.
3. Contraindication to regional anesthesia (coagulopathy, patient refusal).
4. Allergy to local anesthetic or other study medications.
5. BMI > 35 kg/m2.
6. Chronic opioid use (daily or almost daily use for > 3 months).
7. Active illicit drug use.
8. Additional surgical site other than the limb for adductor canal block.
9. Pregnancy.
10. Preexisting neuropathy in the operative limb.
11. Inability to communicate to investigators or hospital staff.
12. Inability to speak or understand English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Missair, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Pressure: High pressure injection of Ropivacaine local anesthetic at greater than 20 psi
  High Pressure Injection: Adductor canal block performed at greater than 20 psi injection pressure
  High Pressure Injection: Ropivacaine 0.2% injection at greater than 20 psi injection pressure
- Low Pressure: Low pressure injection of Ropivacaine local anesthetic at less than 15 psi
  Low Pressure Injection: Adductor canal block performed at less than 15 psi injection pressure
  Low Pressure Injection: Ropivacaine 0.2% injection at less than 15 psi injection pressure
Period: Overall Study
Arm/Group | High Pressure | Low Pressure
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Pressure | Low Pressure | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 5 | 10 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Spread of Injectate
Description: Our primary endpoint is the spread of injectate, defined as the distance between the uppermost and lowermost limits of spread of local anesthetic as assessed by ultrasound.
Time Frame: Immediate post-procedure on day 1
Measure: Mean (Full Range); unit: cm
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
cm | 18.5 [8.5 to 29] | 10 [2 to 16.5]

2. Secondary Outcome: Number of Events of Femoral Nerve Block 30 Minutes After Block Placement
Description: Sensory testing will use a pinprick method in the femoral (anterior thigh), saphenous (medial calf proximal to the medial malleolus, top of the patella) and sciatic (posterolateral calf, plantar surface of the foot) nerve distributions; if patients are unable to feel the stimulus in the femoral nerve distribution, then an outcome of a femoral nerve block will be recorded.
Time Frame: post-procedure and postoperative on day 1
Measure: Number; unit: Events
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
Events | 0 | 0

3. Secondary Outcome: Number of Events of Sciatic Nerve Block 30 Minutes After Block Placement
Description: Sensory testing will use a pinprick method in the femoral (anterior thigh), saphenous (medial calf proximal to the medial malleolus, top of the patella) and sciatic (posterolateral calf, plantar surface of the foot) nerve distributions; if patients are unable to feel the stimulus in the sciatic nerve distribution, then an outcome of a sciatic nerve block will be recorded.
Time Frame: post-procedure and postoperative on day 1
Measure: Number; unit: Events
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
Events | 0 | 0

4. Secondary Outcome: Postoperative Pain Scores (Numeric Rating Scale, 0-10)
Description: Patients will rate their pain after surgery on a scale from 0-10, with 0 being no pain, and 10 being the worst pain of their life.
Time Frame: postoperative on day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
score on a scale | 3 [2 to 3] | 4 [3.25 to 5.75]

5. Secondary Outcome: Postoperative Physical Therapy Milestone Achievement
Description: The patient will be evaluated by physical therapy postoperatively using the Lower Extremity Function Scale (LEFS). The LEFS is a self-reporting measure (0-80 score range, where 0 is complete disability and 80 is fully functional).
Time Frame: postoperative week 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
score on a scale | 47 [18 to 68] | 30 [8 to 55]

6. Secondary Outcome: Postoperative Physical Therapy Milestone Achievement
Description: as for outcome 5
Time Frame: postoperative week 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
score on a scale | 53 [32 to 75] | 50 [22 to 58]

7. Secondary Outcome: Postoperative Physical Therapy Milestone Achievement
Description: as for outcome 5
Time Frame: postoperative week 3
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
score on a scale | 60 [30 to 72] | 51 [40 to 70]

8. Secondary Outcome: Postoperative Physical Therapy Milestone Achievement
Description: as for outcome 5
Time Frame: postoperative week 4
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
score on a scale | 70 [59 to 78] | 65 [20 to 69]

9. Secondary Outcome: Opioid Administration
Description: Intraoperative and immediate postoperative opioid administration. Calculated as morphine milliequivalent (in milligrams).
Time Frame: day 1
Measure: Mean (Standard Error); unit: milligrams
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 12 | 14
milligrams | 20.909 (2.827) | 16.033 (2.438)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Adverse events collected as related to intervention only, as assessed by treating physician.
Arm/Group | High Pressure | Low Pressure
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

LIMITATIONS AND CAVEATS:
Trial was terminated early due to inability to recruit additional subjects after the participating surgeons were staffed at a different hospital and no replacement surgical service was established.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT02563990/Prot_SAP_000.pdf